CLINICAL TRIAL: NCT04961632
Title: An Open-label, Single-institution, Dose-determining (Part 1) and Dose-confirmatory (Part II) Study to Investigate the Optimal Dose of Tamoxifen in Breast Cancer Patients Harboring Different TCF20 rs932376 Variant Alleles
Brief Title: Dose-determining and Dose-confirmatory Study to Investigate the Optimal Dose of Tamoxifen in Breast Cancer Patients According to Genotype Status of TCF20 rs932376
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Cancer Centre, Singapore (Other)
Collaborators: National Medical Research Council (NMRC), Singapore (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TCF20-BRE-01
Record Dates: First submitted 2021-07-05; First posted 2021-07-14 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Tamoxifen

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dose-determination (Experimental)
  Interventions: Drug: Tamoxifen
- Dose-confirmation (Experimental)
  Interventions: Drug: Tamoxifen

INTERVENTIONS:
Drug: Tamoxifen — Patients taking 20mg tamoxifen will receive dose increments of 10mg every 8 weeks until endoxin threshold of >30nM or the maximum dose of 40mg/day is reached. The escalated dose will be taken for 1 year before reverting back to 20mg.
  Arms: Dose-determination
Drug: Tamoxifen — Patients will take tamoxifen at the ascribed genotype-determined dose as determined in the dose-determination phase.
  Arms: Dose-confirmation

SUMMARY:
The investigators hypothesize that the TCF20 rs932376 locus controls endoxifen levels in estrogen receptor (ER)-positive breast cancer patients on tamoxifen therapy and that the requirement of tamoxifen dose to achieve therapeutic levels of endoxifen varies according to the genotype status of the patient's at the TCF20 rs932376 locus.

Patients will receive escalating doses of tamoxifen according to their TCF20 rs932376 genotype status. Patients on 20mg tamoxifen daily for 8 weeks or longer will provide blood samples for analysis of tamoxifen and its metabolites. Patients assess with >30nM endoxifen concentrations will continue with 20mg tamoxifen dose. Patients who have endoxifen concentrations <30nM will receive dose increments of 10mg every 8 weeks until they achieve endoxifen threshold of >30nM or reach maximum dose level of 40mg/day.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed stage I to IV breast cancer
* Age greater than 21 years
* Estrogen- or progesterone-receptor positive tumours
* Patients receiving tamoxifen 20mg daily as monotherapy
* Patients currently taking tamoxifen in either adjuvant or metastatic setting for greater than or equal to 8 weeks (for Dose determination and confirmation phases)
* Patients who will commence on tamoxifen therapy in either adjuvant or metastatic setting (for Dose confirmation phase only)
* Written and informed consent from participating patients

Exclusion Criteria:

* Patients with expected survival less than 6 months
* Patients who are human epidermal growth factor receptor 2 (HER2)-postitive
* Inability to provide informed consent
* Patients receiving CYP2D6 inhibitors or inducers within the past four weeks from the time of study enrollment. However, patients started in CYP2D6 inhibitors or inducers after commencing on tamoxifen therapy will not be excluded from the study.
* Pregnancy
* Patients with prior malignancies other than those who have received curative treatment for basal cell carcinoma of the skin or carcinoma in situ of the uterine cervix
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/ social situations that would limit compliance with study requirements.
* Patients who have documented prior allergic reaction to tamoxifen

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2020-12-23 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Endoxifen blood concentration | 8 weeks after each tamoxifen dose level at 20mg, 30mg and 40mg
  To determine the optimal dose of tamoxifen required to achieve therapeutic endoxifen levels for each TCF20 rs932376 genotype group in the dose-determination phase

CONTACTS AND LOCATIONS:
Overall Officials: Elaine Lim, Principal Investigator — National Cancer Centre, Singapore
Locations (1):
- National Cancer Centre, Singapore, Singapore